CLINICAL TRIAL: NCT03035305
Title: Seasonal Malaria Chemoprevention With or Without Lipid-based Nutrient Supplement in Children Aged 6-59 Months in Kolokani Circle, Koulikoro Region, Mali, August-November 2016: Interventional Matched-pair Clustered Cohort
Brief Title: Seasonal Malaria Chemoprevention With or Without Lipid-based Nutrient Supplement in Children Aged 6-59 Months in Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Alliance médicale contre le paludisme, Mali (Unknown); Programme national de lutte contre le paludisme, Mali (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); European Commission (Other); Ministry of health, Mali (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMC LNS Mali
Record Dates: First submitted 2017-01-17; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Seasonal malaria chemoprevention; Lipid-based nutrient supplement; Children; Mali
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMC and LNS (intervention group) (Experimental): Children included in the 9 health areas of the intervention group receiving both lipid-based nutrient supplement and seasonal malaria chemoprevention with sulfadoxine-pyrimethamine plus amodiaquine
  Interventions: Dietary Supplement: Lipid-based Nutrient Supplement (LNS); Drug: Seasonal malaria chemoprevention
- SMC only (control group) (Other): Children included in the 9 health areas of the control group receiving seasonal malaria chemoprevention with sulfadoxine-pyrimethamine plus amodiaquine
  Interventions: Drug: Seasonal malaria chemoprevention

INTERVENTIONS:
Dietary Supplement: Lipid-based Nutrient Supplement (LNS) — For each round of SMC distribution (total of 4 rounds):
  * For children aged 6-11 months: 15 sachets/month or 50g every two days for 4 weeks
  * For children aged 12-59 months: 21 sachets/month or 50g per day for 3 weeks
  Arms: SMC and LNS (intervention group)
Drug: Seasonal malaria chemoprevention — For each round of SMC distribution (total of 4 rounds):
  * For children aged 6-11 months: sulfadoxine 250mg/pyrimethamine 12.5mg and amodiaquine 75mg
  * For children aged 12-59 months: sulfadoxine 500mg/pyrimethamine 25mg and amodiaquine 150mg
  D1 : 1 tablet sulfadoxine-pyrimethamine + 1 tablet amodiaquine D2 : 1 tablet amodiaquine D3 : 1 tablet amodiaquine
  Other Names: Sulfadoxine-pyrimethamine plus amodiaquine

SUMMARY:
SMC LNS Mali is a interventional matched-pair clustered cohort carried out between August and November 2017 in 18 health areas in Kolokani Circle, Koulikoro region, Mali.

The objective of this study is to determine whether the association SMC and LNS reduces the number of confirmed malaria cases among children 6-59 months during the monthly SMC distribution sessions.

DETAILED DESCRIPTION:
Main objective:

To compare confirmed cases of malaria among children aged 6-59 months between the group receiving SMC combined with LNS (intervention group) and the group receiving only SMC (control group) during the monthly SMC distribution sessions (4 rounds)

Secondary objectives:

To compare among children aged 6-59 months between two groups

* Fever cases
* Acute malnutrition cases (global, moderate and severe)
* Medical referral cases and their reasons

Study site:

The study is conducted in 18 health areas in Kolokani Circle, Koulikoro region, Mali. Each group (intervention and control groups) is composed of 9 health areas.

Number of participants:

Between 17500 and 22000 in each group (estimation)

ELIGIBILITY:
Inclusion Criteria:

* Being between 6 and 59 months old
* Resident in the study area
* Signed informed consent of the mother or the child's guardian

Exclusion Criteria:

* Children allergic to milk, peanuts, sulfadoxine-pyrimethamine or amodiaquine

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36717 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Confirmed malaria case | From the 2nd round of SMC distribution (4 weeks after the date of inclusion) to the 4th round of SMC distribution (12 weeks after the date of inclusion), assessed up to 8 weeks
  Malaria case is confirmed by a positive malaria rapid diagnostic test. This outcome will be defined as the occurrence of at least one confirmed malaria case from the 2nd through the 4th round of SMC distribution.

SECONDARY OUTCOMES:
Fever case | From the 2nd round of SMC distribution (4 weeks after the date of inclusion) to the 4th round of SMC distribution (12 weeks after the date of inclusion), assessed up to 8 weeks
  Fever case is defined by an axillary temperature greater than 37.5⁰C measured by electronic thermometer or notion fever within 48 hours. This outcome will be defined as the occurrence of at least one fever case from the 2nd through the 4th round of SMC distribution.
Global acute malnutrition case | From the 2nd round of SMC distribution (4 weeks after the date of inclusion) to the 4th round of SMC distribution (12 weeks after the date of inclusion), assessed up to 8 weeks
  Global acute malnutrition is defined by MUAC <125mm (orange or red color MUAC) and/or bilateral edema. This outcome will be defined as the occurrence of at least one global acute malnutrition case from the 2nd through the 4th round of SMC distribution.
Moderate acute malnutrition case | From the 2nd round of SMC distribution (4 weeks after the date of inclusion) to the 4th round of SMC distribution (12 weeks after the date of inclusion), assessed up to 8 weeks
  Moderate acute malnutrition is defined by MUAC between 115-124mm (orange color MUAC). This outcome will be defined as the occurrence of at least one moderate acute malnutrition case from the 2nd through the 4th round of SMC distribution.
Severe acute malnutrition case | From the 2nd round of SMC distribution (4 weeks after the date of inclusion) to the 4th round of SMC distribution (12 weeks after the date of inclusion), assessed up to 8 weeks
  Severe acute malnutrition is defined by MUAC <115mm (red color MUAC) and/or bilateral edema. This outcome will be defined as the occurrence of at least one severe acute malnutrition case from the 2nd through the 4th round of SMC distribution.
Medical referral case | From the 2nd round of SMC distribution (4 weeks after the date of inclusion) to the 4th round of SMC distribution (12 weeks after the date of inclusion), assessed up to 8 weeks
  This outcome will be defined as the occurrence of at least one illness of sufficient severity to warrant referral to the nearest medical structure for evaluation from the 2nd through the 4th round of SMC distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shepherd, MD, Principal Investigator — The Alliance for International Medical Action (ALIMA); Renaud Becquet, PhD, Principal Investigator — Inserm U1219 Bordeaux Population Health Center, University of Bordeaux
Locations (1):
- Amcp/Alima, Kolokani Circle, Koulikoro, Mali

IPD SHARING:
Plan to Share IPD: No